CLINICAL TRIAL: NCT05554952
Title: Indirect Pulp Capping Versus Pulpotomy With MTA for Treatment of Primary Molars With Deep Caries: An Equivalent Parallel Randomized Controlled Trial
Brief Title: Indirect Pulp Capping Versus Pulpotomy With MTA for Treatment of Primary Molars With Deep Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hasnaa monis, Resident in pediatric dentistry department faculty of dentistry assuit university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 526_1 /11/2021
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Indirect Pulp Capping; Pulpotomy
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Indirect pulp capping with MTA
  Interventions: Combination Product: MTA
- Group 2 (Active Comparator): Pulpotomy with MTA
  Interventions: Combination Product: MTA

INTERVENTIONS:
Combination Product: MTA — Mineral trioxide aggregate (MTA) is composed of Portland cement, with 4:1 addition of bismuth oxide added so that the material can be detected on a radiograph. The cement is made up of calcium, silicon and aluminium. The main constituent phases are tricalcium and dicalcium silicate and tricalcium aluminate.

SUMMARY:
The aim of the current randomized controlled trial is to evaluate clinical and radiographic outcomes of indirect pulp capping and pulpotomy with MTA in treatment of primary teeth with deep caries over a 12-month follow-up period.

DETAILED DESCRIPTION:
Output patients coming to Pediatric dentistry department Minia University, selected randomly to evaluate clinical and radiographic outcomes of indirect pulp capping and pulpotomy with MTA in treatment of primary teeth with deep caries over a 12-month follow-up period an equivalent parallel randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* - 4 to 6 years old patients presented with deep carious lesions in primary molars.
* Apparently healthy children (ASA I, II classification).
* Co-operative children (Rating 3 & 4 according to Frankle classification)

Exclusion Criteria:

A) Clinical:

* Non restorable primary molars.
* Presence of clinical pathology.
* Presence of mobility or tenderness to percussion.

  * Spontaneous pain.

B) Radiographic:

* Pre-operative radiographs showed external or internal root resorption.
* Presence of furcal radiolucency.
* Presence of periapical radiolucency or widened periodontal ligament space
* More than one-third root resorption detected.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic evaluation | 2 years follow up
  The children will be recalled for postoperative clinical and radiographic assessment at the following intervals: 3, 6, 12 months the treatment will be considered successful if none of the following clinical or radiographic findings is present:
  Clinical criteria:
  1. pain
  2. tenderness to palpation or percussion
  3. gingival swelling or sinus tract
  4. purulent exudate expressed from the gingival margin
  5. abnormal tooth mobility
  Radiographic criteria:
  1. periapical radiolucency
  2. widening in peridontal ligament space

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt